CLINICAL TRIAL: NCT05393674
Title: A Phase II Study of Fedratinib and Nivolumab Combination in Patients With Myelofibrosis and Resistance or Suboptimal Response to JAK-inhibitor Treatment
Brief Title: Fedratinib in Combination With Nivolumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Prof. F. Heidel, MH Hannover (Unknown); Celgene International II S.á.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRACTION_2021
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
Keywords: MF; Fedratinib; JAK-inhibitor; Nivolumab
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Fedratinib (Cycle 1: Run-in-Phase with 400 mg QD for 4 weeks, Cycle 2-12: 400 mg QD, Dose modifications will be allowed based on observed toxicity to a 300 mg or a 200 mg daily dose) + Nivolumab (Cycle 2-12: 240 mg, i.v., q2w)
  Patients will receive study treatment until loss of response, death or study discontinuation for other reasons.
  Interventions: Drug: Fedratinib Oral Capsule [Inrebic]; Drug: Nivolumab

INTERVENTIONS:
Drug: Fedratinib Oral Capsule [Inrebic] — 400 mg once daily p.o. from cycle 1-n, dose adjustment will be made according to the protocol
Drug: Nivolumab — 240 mg every 2 weeks i.v. from cycle 2-n

SUMMARY:
A multicenter, open-label, single arm, phase II study investigating the clinical efficacy of Fedratinib and Nivolumab combination in patients with myelofibrosis and resistance or suboptimal response to JAK-inhibitor treatment

DETAILED DESCRIPTION:
The FRACTION trial will evaluate the clinical efficacy of Fedratinib and Nivolumab combination therapy in patients with primary and secondary myelofibrosis based on the consensus criteria of the International Working Group for Myelofibrosis Research and treatment (IWG-MRT), extended by the criterion RBC-transfusion independence (RBC-TI).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form available and patient willing and able to adhere to the study visit schedule and other protocol requirements.
2. Patients* ≥18 years of age
3. diagnosed with myelofibrosis (MF) according to the WHO 2008 or 2016 criteria, including primary (pre-fibrotic or overt) and secondary myelofibrosis.
4. Patients with an indication for therapy (either symptomatic patients with splenomegaly >11cm diameter and/or symptoms restricting their daily activity or patients with DIPSS int-2, or high risk or MIPSS70 int or high)
5. Patients with no response or suboptimal response to any JAK-inhibitor therapy (regarding persistence of symptoms, splenomegaly, cytopenia or hyperproliferation) defined either by

   * Persisting Splenomegaly >11cm total diameter
   * OR Persisting leukoerythroblastosis
   * OR Anemia <6.2 mmol/l (<10g/dl)
   * OR Elevated WBC (>11 Gpt/l)
   * OR Persisting general or constitutional symptoms (persistence is defined as less than 50% reduction to baseline when using the MPN10 TSS Score)
   * OR failure [secondary resistance] to JAK-inhibitor treatment as defined by IWG-MRT criteria.
6. ECOG performance status <3 at screening and adequate organ function
7. Reliable contraception should be maintained throughout the study and for 1 month after discontinuation of Fedratinib or 5 months after discontinuation of Nivolumab**
8. Subject must be willing to receive transfusion of blood products
9. Thiamine levels not below lower limit of normal (prior substitution is possible)
10. Normal nutritional status, as judged by the physician
11. Females of childbearing potential (FCBP) must undergo repetitive pregnancy testing (serum or urine) and pregnancy results must be negative.
12. Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods (i.e. failure rate of < 1% per year).
13. Males (including those who have had a vasectomy) must use barrier contraception (condoms) when engaging in sexual activity with FCBP. Males must agree not to donate semen or sperm.

Exclusion Criteria:

1. Planned hematopoietic stem cell transplantation within 3 months and suitable donor available
2. >10% blasts in bone marrow smear (cytology) or >2x in blood smear within the screening phase or >20% blasts at any time in bone marrow or peripheral blood smears
3. Creatinine >2xULN and Creatinine-Clearance <45ml/min; ALAT, ASAT & bilirubin >3xULN (if MF impact on liver >5xULN)
4. Baseline platelets count below 50 x 10^9/L and ANC < 1.0 x 10^9/L
5. Diagnosis of PV, ET (according to WHO 2016) or positive molecular test for BCR-ABL
6. Patients on ongoing medication for myelofibrosis including systemic corticosteroids (detailed list of permitted medications is provided in paragraph 9.1.10.4 and Appendix V). Use of steroids within 14 days prior to the first dose of study drug and until end of treatment is prohibited by patients.
7. Uncontrolled infection
8. Evidence of acute or chronic infection with hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or tuberculosis
9. Current participation in any other interventional clinical study within 30 days before the first administration of the investigational product or at any time during the study, unless it is an observational (non-interventional) study, or during the follow-up period of an interventional study with last dose of investigational product ≥30 days prior first administration of investigational product within this study.
10. No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician about study participation
11. No consent for biobanking of patient's biological specimens
12. Prior therapy with checkpoint-inhibitors
13. Vaccination within 4 weeks prior to treatment start
14. Hypersensitivity to the IMPs or to any of the excipients
15. History of or uncontrolled autoimmune disease such as autoimmune-hepatitis, -pneumonitis, -thyroiditis, chronic inflammatory bowel disease, multiple sclerosis, or rheumatologic diseases (including but not limited to systemic lupus and vasculitis)
16. History of malignancy except for i) adequately treated local basal cell or squamous cell carcinoma of the skin, ii) asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to randomization, or iii) any other cancer that has been in complete remission for ≥ 5 years
17. Secondary malignancy that limits survival to less than 6 months.
18. Drug or alcohol abuse within the last 6 months
19. Patients who cannot adhere to the Pregnancy Prevention Plan
20. Pregnant or breast-feeding females
21. Thiamine levels below normal limit despite supplementation
22. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Best response rate within 12 treatment cycles | 12 months after therapy start.
  Best response rate within 12 treatment cycles according to the IWG-MRT criteria (including complete remission, CR, partial remission, PR, clinical improvement, CI, stable disease, SD 1, and red cell transfusion (RCT) independency according to Gale et al.)

SECONDARY OUTCOMES:
Safety: Incidence and severity of adverse events according to CTC criteria | From informed consent until 100 days after last study drug
  Incidence and severity of adverse events according to CTC criteria
Safety: Timing of adverse events according to CTC criteria | From informed consent until 100 days after last study drug
  Timing of adverse events according to CTC criteria
Safety: Incidence of Laboratory abnormalities | From informed consent until 100 days after last study drug
  Incidence of laboratory abnormalities including timing and relatedness.
Safety: leukemic transformation | From informed consent until 100 days after last study drug
  Cumulative incidence of leukemic transformation
Clinical benefit | 3.5 years
  Proportion of patients with clinical benefit defined as stable disease (SD) plus hematologic improvement or stable disease (SD) plus improvement of MF-associated symptoms
Efficacy: PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 42 months
  Progression-free survival
Efficacy: Duration of response | 3.5 years
  Time from first response including RBC-TI, CI, PR and CR (Appendix III) to date of loss of response. Times of patients without loss of response are censored at last tumor assessment.
Efficacy: Overall survival | 3.5 years
  Time from study entry to the last date known to be alive or death. Survival times of patients alive at last follow-up are censored.
Efficacy: Disease burden | 3.5 years
  Change of disease burden assessed by allelic ratio of the respective driver mutation and of high-risk mutations by next-generation sequencing [NGS]

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH
Locations (7):
- Germany (7):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - University Medicine Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - Medizinische Hochschule, Hanover
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Johannes Wesling Klinikum, Minden
  - Uniklinik Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Result] Isfort S, von Bubnoff N, Al-Ali HK, Becker H, Gotze T, le Coutre P, Griesshammer M, Moskwa C, Wohn L, Riedel J, Palandri F, Manz K, Hochhaus A, Dohner K, Heidel FH. FRACTION: protocol of a phase II study of Fedratinib and Nivolumab combination in patients with myelofibrosis and resistance or suboptimal response to JAK-inhibitor treatment of the German MPN study group (GSG-MPN). Ann Hematol. 2024 Aug;103(8):2775-2785. doi: 10.1007/s00277-024-05867-w. Epub 2024 Jul 5. PMID 38967662